CLINICAL TRIAL: NCT03977662
Title: Pancreatic Islets and Parathyroid Gland Co-transplantation for Treatment of Diabetes in the Intra-Muscular Site
Brief Title: Pancreatic Islets and Parathyroid Gland Co-transplantation for Treatment of Type 1 Diabetes
Acronym: PARADIGM
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Peter Stock (Other)
Collaborators: California Institute for Regenerative Medicine (CIRM) (Other)
Responsible Party: Sponsor-Investigator, Peter Stock, Principle Investigator, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-26725
Record Dates: First submitted 2019-05-24; First posted 2019-06-06 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PTG with adult pancreatic islet co-transplantation (Experimental): People with Type 1 (c-peptide negative) diabetes with stable kidney or liver allografts on chronic immunosuppression who receive study intervention, which is co-transplantation of allogeneic parathyroid (PTG) with adult pancreatic islets in people with Type 1 diabetes in the intramuscular (IM) site
  Interventions: Combination Product: Co-transplantation of PTG with pancreatic islets

INTERVENTIONS:
Combination Product: Co-transplantation of PTG with pancreatic islets — Co-transplantation of allogeneic parathyroid glands (PTG) with adult pancreatic islets (both PTG and pancreatic islets obtained from same deceased donor) in people with Type 1 diabetes in the intramuscular (IM) site with stable function of liver or kidney allografts on chronic immunosuppression

SUMMARY:
The primary objective is to test the hypothesis that co-transplantation of allogeneic PTG with adult pancreatic islets (derived from same deceased donor) in the IM site in people with Type 1 diabetes with functioning kidney and/or liver transplants is safe, allows islet engraftment, and leads to insulin independence.

DETAILED DESCRIPTION:
Single-center, open label, non-randomized safety and efficacy trial to evaluate co-transplantation of allogeneic parathyroid glands (PTG) with adult pancreatic islets (both PTG and pancreatic islets obtained from same deceased donor) in people with Type 1 diabetes in the intramuscular (IM) site with stable function of liver or kidney allografts on chronic immunosuppression.

A total of 8 patients will be enrolled in the study and followed for a minimum of 1 year up to 2 years after the last islet transplant, depending on enrollment date.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects age 18 or older.
2. Subjects who are able to provide written informed consent and to comply with study procedures.
3. Clinical history compatible with Type 1 diabetes (onset < 40 yrs old and insulin dependent for > 5 yrs at enrollment, c-peptide negative).
4. Recipients should have absent stimulated c-peptide (< 0.3 ng/mL) in response to a (Boost® 6 mL/kg BW to a maximum of 360 mL; another equivalent product), measured at 60 and 90 min after start of consumption.
5. Subjects who are > 6 months post-renal transplant or >6 months post-liver transplant who are taking appropriate calcineurin inhibitor (CNI) based maintenance immunosuppression ([tacrolimus alone or in conjunction with sirolimus, mycophenolate mofetil, myfortic, or azathioprine; or cyclosporine in conjunction with sirolimus, mycophenolate mofetil, or myfortic ± Prednisone ≤ 10 mg/day).
6. Stable renal function as defined by a creatinine of no more than one third greater than the average creatinine determination performed in the 6 previous months prior to islet transplant, as well as absence of a rejection episode in the 6 months prior to islet transplant
7. Stable liver function tests as defined by: SGOT (AST), SGPT (ALT), alkaline phosphatase values < 1.5, or total bilirubin < 1.5 times normal upper limits at time of study entry, as well as absence of a rejection episode in the 6 months prior to islet transplant

Exclusion Criteria:

1. Presence of donor specific anti-HLA antibodies detected by Luminex Single Antigen/specificity bead assay including weakly reactive antibodies that would not be detected by a flow cross match
2. Insulin requirement of >1.0 IU/kg/day
3. Weight more than 100 kg or body mass index (BMI) > 30 kg/m2.
4. Primary hyperparathyroidism OR secondary hyperparathyroidism
5. Untreated or unstable proliferative diabetic retinopathy.
6. Blood Pressure: SBP > 180 mmHg or DBP >100 mmHg despite treatment with antihypertensive agents.
7. Calculated GFR of ≤ 40 mL/min/1.73 m2 using the subject's measured serum creatinine and the Chronic Kidney Disease Epidemiology Collaboration (CKD- EPI) equation, as well as presence of a rejection episode in the 6 months prior to islet transplant
8. Elevated liver function tests as defined by: SGOT (AST), SGPT (ALT), alkaline phosphatase values > 1.5, or total bilirubin >1.5 times normal upper limits at time of study entry, as well as presence of a rejection episode in the 6 months prior to islet transplant
9. Proteinuria (albumin/creatinine ratio or ACr > 300mg/g) of new onset since kidney transplantation.
10. For female subjects: Positive pregnancy test, presently breast-feeding, or unwillingness to use effective contraceptive measures for the duration of the study and 4 months after discontinuation. For male subjects: intent to procreate during the duration of the study or within 4 months after discontinuation or unwillingness to use effective measures of contraception. Oral contraceptives, Norplant®, Depo- Provera®, and barrier devices with spermicide are acceptable contraceptive methods; condoms used alone are not acceptable.
11. Active infection including hepatitis B, hepatitis C, HIV, or TB. Quantiferon gold assay will be used to determine TB infection.
12. Invasive aspergillus, histoplasmosis, and coccidioidomycosis infection within 1 year prior to study entry.
13. Any history of malignancy following receiving either the kidney or liver transplant, except for completely resected squamous or basal cell carcinoma of the skin
14. Known active alcohol or substance abuse.
15. Severe co-existing cardiac disease, characterized by any one of these conditions:

    1. Recent MI (within past 6 months),
    2. Evidence of ischemia on functional cardiac exam within the last year,
    3. Left ventricular ejection fraction < 30%,
    4. Valvular disease requiring replacement with prosthetic valve.
16. Active infections (except mild skin and nail fungal infections).
17. Use of any investigational agents within 4 weeks of enrollment.
18. Administration of live attenuated vaccine(s) within 2 months of enrollment.
19. Any medical condition that, in the opinion of the investigator, will interfere with safe study completion.
20. Positive screen for BK viremia at time of screening.
21. Untreated hyperlipidemia - TC > 200 mg/dL, TGC > 200 mg/dL, LDL > 130 mg/dL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Minimum of 1 year up to 2 years depending on transplant date
  Safety: Since this study is a pilot non-randomized safety and efficacy trial with patient enrollment limited by budgetary constraints, no direct statistical significance tests can be performed.
Incidence of post-transplant infections and malignancies | Minimum of 1 year up to 2 years depending on transplant date
  Safety: Since this study is a pilot non-randomized safety and efficacy trial with patient enrollment limited by budgetary constraints, no direct statistical significance tests can be performed.
Incidence of de novo sensitization | Minimum of 1 year up to 2 years depending on transplant date
  Safety: Since this study is a pilot non-randomized safety and efficacy trial with patient enrollment limited by budgetary constraints, no direct statistical significance tests can be performed.
Incidence of Insulin independence | Minimum of 1 year up to 2 years depending on transplant date
  Efficacy: Incidence of participants no longer using insulin

SECONDARY OUTCOMES:
Glycemic control | Day 75, Day 180, Day 270, Year 1, Year 1.5, Year 2
  Assessed by measuring HbA1c using high-performance liquid chromatography
Hypoglylcemic episodes: Clarke Survey Score | Day 75, Day 180, Day 270, Year 1
  The Clarke survey will be used to assess the frequency and severity of hypoglycemic episodes
Hypoglylcemic episodes: Hypo Score | Day 75, Day 180, Day 270, Year 1
  The HYPO score will be used to assess the frequency and severity of hypoglycemic episodes
Beta cell function as assessed by Mixed Meal Tolerance Test (MMTT) | Day 75, Day 180, Day 270, Year 1, Year 1.5, Year 2
  Results from both MMTT and FSIGT will be used to assess beta cell function
Beta cell function as assessed by Insulin-Modified Frequently-Sampled Intravenous Glucose ToleranceTest (FSIGT) | Day 75, Day 180, Day 270, Year 1, Year 1.5, Year 2
  Results from both MMTT and FSIGT will be used to assess beta cell function

CONTACTS AND LOCATIONS:
Overall Officials: Peter Stock, MD, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, California, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-20): https://cdn.clinicaltrials.gov/large-docs/62/NCT03977662/Prot_SAP_002.pdf